CLINICAL TRIAL: NCT01835873
Title: Comparative Study of the Effect of 6% Hydroxyethyl Starch 130/0.42 vs Lactated Ringer's Preload on the Hemodynamic Status of Parturients Undergoing Spinal Anesthesia for Elective Cesarean Delivery. Arterial Pulse Contour Analysis (FloTrac/VigileoTM) is Employed for Continuous Monitoring of Maternal Hemodynamic Parameters
Brief Title: The Effect of Intravenous Prehydration on the Hemodynamic Status of Healthy Parturients Undergoing Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paraskevi Matsota (Other)
Responsible Party: Sponsor-Investigator, Paraskevi Matsota, Assistant Professor of Anesthesiology, MD, PhD, Attikon Hospital
Organization: Attikon Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 492
Record Dates: First submitted 2013-04-06; First posted 2013-04-19 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Ringer's Lactate; HES 130-0.42-6:1

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lactated Ringer's (Active Comparator): Crystalloid solution - 1000 ml preload
  Interventions: Other: Lactated Ringer's
- HES 130/0.42 (Active Comparator): Hydroxyethyl starch (HES 130/0.42) - 500 ml preload
  Interventions: Other: HES 130/0.42

INTERVENTIONS:
Other: Lactated Ringer's
  Arms: Lactated Ringer's
Other: HES 130/0.42 — Balanced colloid solution
  Other Names: Tetraspan® 6%
  Arms: HES 130/0.42

SUMMARY:
Regional anesthesia (spinal, epidural) is considered the method of choice for anesthesia obstetric deliveries because of the ability to use fewer drugs, a more direct experience of childbirth and the capability to provide excellent postoperative analgesia. However, the incidence of hypotension after spinal anesthesia for cesarean delivery is high and can lead to maternal and fetal morbidities. Certain interventions may reduce the incidence and severity of spinal anesthesia induced hypotension, including the use of vasopressors and intravenous pre- or co-hydration using different types of volume expanders; crystalloid or colloid solutions. Such interventions aim to increase maternal cardiac output, which is the key in attenuating the hypotensive response to spinal anesthesia.

The primary purpose of this study is to compare the efficacy of intravenous prehydration (preloading) of healthy parturients scheduled for caesarean section with either a crystalloid (Ringer's lactated) or colloid solution (HES 130/0.42) in the prevention of hypotension after spinal anesthesia.

The FloTrac/VigileoTM device provides continuous monitoring of maternal cardiac output by employment of a minimally invasive technique based on arterial pulse contour analysis. Assessment of maternal hemodynamic status using the FloTrac/VigileoTM constitutes a secondary outcome. Other secondary outcomes are total amount of vasopressors used, neonatal outcome, intraoperative side effects and maternal satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I and II parturients
* singleton gestation
* term gestation (gestational period more than 37 weeks)

Exclusion Criteria:

* extremes of weight (<50 Kgr or >120 Kgr)
* extremes of height (<150 cm or >180 cm)
* baseline heart rate less than 65 bpm
* active labor
* known fetal abnormalities
* placental abruption, placenta previa/accreta
* pregnancy induced hypertension
* anemia (hemoglobin < 9 gr/dl)
* cardiac, respiratory or renal disease
* diabetes mellitus
* spinal cord abnormalities
* previous spinal surgery
* preexisting neurological dysfunction
* known allergy to any protocol medication
* any absolute contraindication to regional anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of spinal anesthesia induced hypotension in elective cesarean deliveries preloaded with either crystalloid or colloid solution. | Maternal hemodynamic data is assessed before volume preload, immediately after volume preload, immediately after spinal anesthesia and at one minute intervals thereafter until placental delivery. Expected average of 40 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece